CLINICAL TRIAL: NCT04041050
Title: A Phase 1 Open-Label Study Evaluating the Safety and Tolerability, and Pharmacokinetics of Navitoclax Monotherapy and in Combination With Ruxolitinib in Myeloproliferative Neoplasm Subjects
Brief Title: A Study Evaluating Safety and Tolerability, and Pharmacokinetics of Navitoclax Monotherapy and in Combination With Ruxolitinib in Participants With Myeloproliferative Neoplasm
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M19-753; 2020-002597-27 (EudraCT Number)
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-06

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Myeloproliferative Neoplasm (MPN); Chronic myelomonocytic leukemia (CMML); Polycythemia Vera (PV); Essential Thrombocythemia (ET); Myelofibrosis (MF); cancer; navitoclax; ruxolitinib
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Neoplasms | interventions — navitoclax; ruxolitinib; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1: Navitoclax Monotherapy (Experimental): Participants will receive various doses of navitoclax once daily (QD).
  Interventions: Drug: Navitoclax
- Part 2: Navitoclax + Ruxolitinib Combination Therapy (Experimental): Participants will receive various doses of navitoclax once daily (QD) in combination with ruxolitinib twice daily (BID).
  Interventions: Drug: Navitoclax; Drug: Ruxolitinib
- Part 3: Navitoclax Monotherapy (Experimental): Participants will receive navitoclax once daily (QD).
  Interventions: Drug: Navitoclax
- Part 4: Navitoclax + Celecoxib (Experimental): Participants will receive navitoclax once daily (QD) starting on Day 3. Participants will also receive celecoxib single dose on Day 1 and Day 7.
  Interventions: Drug: Navitoclax; Drug: Celecoxib
- Part 5: Navitoclax + Ruxolitinib Combination Therapy (Experimental): Participants will receive ruxolitinib BID and navitoclax QD for drug-drug interaction (DDI) assessment, followed by continued administration of navitoclax in combination with ruxolitinib.
  Interventions: Drug: Navitoclax; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Navitoclax — Tablet; Oral
  Other Names: ABT-263
Drug: Ruxolitinib — Tablet; Oral
  Arms: Part 2: Navitoclax + Ruxolitinib Combination Therapy; Part 5: Navitoclax + Ruxolitinib Combination Therapy
Drug: Celecoxib — Capsule; Oral
  Other Names: Celebrex
  Arms: Part 4: Navitoclax + Celecoxib

SUMMARY:
There are 5 parts to this study for which the primary objectives are to evaluate safety, tolerability, and pharmacokinetics (PK) of navitoclax when administered alone (Part 1) or when administered in combination with ruxolitinib (Part 2). In Part 2, participants must have been receiving a stable dose of ruxolitinib therapy for at least 12 weeks prior to study enrollment. In Part 3, all eligible participants will receive navitoclax, with the primary objective being to evaluate potential navitoclax effect on QTc prolongation. In Part 4, effect of navitoclax is evaluated on the PK, safety, and tolerability of a single dose of celecoxib. In Part 5, all eligible participants will receive ruxolitinib twice daily and navitoclax once daily for drug-drug interaction (DDI) assessment, followed by continued administration of navitoclax in combination with ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

Parts 1 and 2:

* Navitoclax Monotherapy (Part 1 Only - Japanese Participants):

  * Documented diagnosis of myelofibrosis (MF), polycythemia vera (PV) or essential thrombocythemia (ET) as defined by the World Health Organization (WHO) classification.
  * MF participants must have received and failed or are intolerant to ruxolitinib therapy.
  * ET or PV participants must be requiring cytoreduction who have failed or are intolerant to at least one prior therapy, or who refuse standard therapy.
* Navitoclax + ruxolitinib Combination Therapy (Part 2 Only - Japanese and Taiwanese Participants):

  * Has documented diagnosis of primary MF, post-polycythemia vera MF (PPV-MF), or post-essential thrombocythemia (PET-MF) as defined by the World Health Organization (WHO) classification.
  * Is ineligible or unwilling to undergo stem cell transplantation at time of study entry.
  * Has splenomegaly as defined by a spleen palpable >= 5 cm below costal margin or spleen volume >= 450 cm^3 as assessed by magnetic resonance imaging (MRI) or computed topography (CT) scan.
  * Must have received ruxolitinib therapy for at least 12 weeks and be currently on a stable dose of ruxolitinib (as described in the protocol).
* Must have adequate bone marrow, kidney, liver and hematology blood values as detailed in the study protocol.
* Part 1 only: Cytoreduction for participants with ET and PV therapy within 14 days prior to the first dose of navitoclax will be allowed pending additional discussion with study doctor. Ruxolitinib for MF participants will not be allowed within 7 days prior to the first dose of study drug and during navitoclax administration.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1.

Part 3, and Part 4 (Participants in US and Europe):

* Part 3 Only: At screening or baseline (pre-dose on Day 1), participant has QT interval corrected for heart rate (QTc) interval by Fridericia's correction (QTcF) <= 450 msec.
* Participants with a documented diagnosis of primary or secondary MF, ET, PV or chronic myelomonocytic leukemia (CMML) as defined by the WHO classification.
* Participants must be requiring treatment and have failed or are intolerant to at least one prior therapy or who refuse standard therapy.
* ECOG performance status <= 2.
* Must have adequate bone marrow, kidney, liver and hematology blood values as detailed in the study protocol.

Part 5 (Participants in US and Europe):

* Has a documented diagnosis of primary MF as defined by the WHO classification, post-polycythemia vera (PV) MF, or post-essential thrombocythemia (ET) MF.
* Classified as intermediate-2 or high-risk MF, as defined by the Dynamic International Prognostic Scoring System (DIPSS).
* Requiring treatment for MF and must either have no prior treatment with a JAK2 inhibitor or have received treatment with ruxolitinib as noted in the protocol.
* Have an ECOG performance status <=2.
* Have adequate bone marrow, kidney, liver and hematology blood values as detailed in the protocol.

Exclusion Criteria:

Part 1 and 2:

* Shows leukemic transformation (> 10% blasts in peripheral blood or bone marrow biopsy).
* Has a history of an active malignancy other than MPN within the past 2 years prior to study entry (exceptions detailed in the protocol).
* Has a positive test result for HIV at screening.
* Has chronic active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment.
* Has evidence of other clinically significant uncontrolled condition(s).
* Has previously taken a BH3 mimetic compound.
* Currently on medications that interfere with coagulation (including warfarin) or platelet function with the exception of low dose aspirin (up to 100 mg) and low-molecular-weight heparin (LMWH).
* Has received strong or moderate CYP3A inhibitors (e.g., ketoconazole, clarithromycin) within 14 days prior to the administration of the first dose of navitoclax.

Part 3, and Part 4:

* Had prior therapy with a BH3 mimetic compound.
* Have received strong or moderate CYP3A inhibitors within 28 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of navitoclax.
* Have received strong CYP3A inducers within 10 days prior to the first dose of navitoclax.
* Show leukemic transformation (> 10% blasts in peripheral blood or bone marrow biopsy).
* Currently on medications that interfere with coagulation (including warfarin) or platelet function except for low-dose aspirin (up to 100 mg) and LMWH.

Part 4 Only:

* Have received CYP2C9 inhibitors within 28 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of study drugs.
* Have received CYP2C9 inducers within 10 days prior to the first dose of study drugs.

Part 5 Only:

* Have accelerated MF, defined as > 10% blasts in peripheral blood or bone marrow aspirate and biopsy.
* Eligible for stem cell transplantation at time of study entry.
* Had prior therapy with a BH3 mimetic compound or BET inhibitor.
* Currently on medications that interfere with coagulation (including warfarin) or platelet function except for low-dose aspirin (up to 100 mg) and LMWH.
* Have received strong CYP3A inhibitors or CYP2C9 inhibitors within 28 days of 5 half-lives of the drug (whichever is shorter) prior to the first dose of study drugs.
* Have received strong CYP3A inducers or CYP2C9 inducers within 10 days prior to the first dose of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLT) (Part 1 and Part 2) | Up to 28 days after the navitoclax initiation
  Dose limiting toxicities for dose escalation purposes will be determined on events that occur during the first 28-day cycle of navitoclax.
Maximum Observed Plasma Concentration (Cmax) of Navitoclax (Part 2 and 5) | Up to approximately 1 day
  Maximum Observed Plasma Concentration (Cmax) of Navitoclax.
Maximum Observed Plasma Concentration (Cmax) of Celecoxib (Part 4) | Up to approximately 1 day
  Maximum Observed Plasma Concentration (Cmax) of Celecoxib.
Time to Cmax (peak time, Tmax) of Navitoclax (Part 2 and 5) | Up to approximately 1 day
  Tmax defined as time to maximum observed plasma concentration of Navitoclax.
Time to Cmax (peak time, Tmax) of Celecoxib (Part 4) | Up to approximately 1 day
  Tmax defined as time to maximum observed plasma concentration of Celecoxib.
Area Under the Plasma Concentration-time Curve from time 0 to the time of the last measurable concentration (AUCt) of Navitoclax | Up to approximately 2 days
  Area under the plasma concentration-time curve from time zero to the last measurable concentration of Navitoclax.
Area Under the Plasma Concentration-time Curve from time 0 to the time of the last measurable concentration (AUCt) of Celecoxib (Part 4) | Up to approximately 2 days
  Area under the plasma concentration-time curve from time zero to the last measurable concentration of Celecoxib.
Number of Participants with Adverse Events | From first dose of study drug until 30 days following last dose of study drug (up to approximately 5 years).
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Change in QT interval corrected for heart rate interval by Fridericia's correction formula (QTcF) (Part 3) | From first dose of study drug until 30 days following last dose of study drug.
  Change in QTcF (Part 3).

SECONDARY OUTCOMES:
Overall Response Rate | Up to approximately 96 weeks
  ORR according to the International Working Group-Myeloproliferative Neoplasms Research and Treatment/European Leukemia Net (IWG-MRT/ELN) criteria for participants with myelofibrosis, essential thrombocythemia, and polycythemia vera, and according to IWG criteria for participants with CMML.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (42):
- United States (12):
  - City of Hope /ID# 239769, Duarte, California
  - Providence - St. Jude Medical Center /ID# 242558, Fullerton, California
  - Moores Cancer Center at UC San Diego /ID# 229584, La Jolla, California
  - UCLA /Id# 222784, Los Angeles, California
  - Northwestern University Feinberg School of Medicine /ID# 224203, Chicago, Illinois
  - Norton Cancer Institute - St. Matthews /ID# 239300, Louisville, Kentucky
  - Duplicate_Brigitte Harris Cancer Pavilion /ID# 238686, Detroit, Michigan
  - Nebraska Cancer Specialists - Omaha - Wright Street /ID# 242554, Omaha, Nebraska
  - Duplicate_East Carolina University Brody School of Medicine /ID# 238560, Greenville, North Carolina
  - Gabrail Cancer Center Research /ID# 228924, Canton, Ohio
  - Pennsylvania Cancer Specialists Research Institute - Gettysburg /ID# 242550, Gettysburg, Pennsylvania
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 228169, Richmond, Virginia
- Cliniques Universitaires UCL Saint-Luc /ID# 225314, Woluwe-Saint-Lambert, Brussels Capital, Belgium
- Bulgaria (2):
  - UMHAT Sveti Georgi /ID# 240022, Plovdiv
  - UMHAT Sveti Ivan Rilski /ID# 240077, Sofia
- Klinicki bolnicki centar Zagreb /ID# 240140, Zagreb, City of Zagreb, Croatia
- France (4):
  - Centre Antoine Lacassagne - Nice /ID# 242293, Nice, Alpes-Maritimes
  - CHU Amiens-Picardie Site Sud /ID# 240792, Amiens, Somme
  - AP-HP - Hopital Saint-Louis /ID# 240685, Paris
  - IUCT Oncopole /ID# 242353, Toulouse
- Germany (4):
  - Universitaetsklinikum Freiburg /ID# 222791, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Kassel /ID# 225440, Kassel, Hesse
  - Universitaetsmedizin Rostock /ID# 225436, Rostock, Mecklenburg-Vorpommern
  - Charite Universitaetsklinikum Berlin - Campus Virchow /ID# 224835, Berlin
- Italy (3):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 221408, Rome, Lazio
  - ASST Spedali civili di Brescia /ID# 224962, Brescia
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRCCS /ID# 224071, Meldola
- Japan (5):
  - Shonan Kamakura General Hospital /ID# 224315, Kamakura-shi, Kanagawa
  - Kindai University Hospital /ID# 213241, Osakasayama-shi, Osaka
  - Osaka University Hospital /ID# 213235, Suita-shi, Osaka
  - Juntendo University Hospital /ID# 213255, Bunkyo-ku, Tokyo
  - University of Yamanashi Hospital /ID# 229279, Chuo-shi, Yamanashi
- University Clinical Center Serbia /ID# 240674, Belgrade, Beograd, Serbia
- Spain (3):
  - Hospital Duran i Reynals /ID# 224007, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra - Pamplona /ID# 224839, Pamplona, Navarre
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 226041, Madrid
- Sweden (2):
  - Duplicate_Karolinska University Hospital /ID# 239992, Stockholm, Stockholm County
  - Linkoping University Hospital /ID# 239995, Linköping
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 215631, Kaohsiung City
  - China Medical University Hospital /ID# 215634, Taichung
- Dokuz Eylul University Medical Faculty /ID# 239952, Izmir, Turkey (Türkiye)
- Gloucestershire Hospitals NHS Foundation Trust /ID# 241189, Cheltenham, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No